CLINICAL TRIAL: NCT05166668
Title: Impact of Adding Letrozole to Gonadotrophin-Releasing Hormone Antagonist Protocol in Women Over 40 Years Undergoing ICSI Cycle
Brief Title: Letrozole /GnRH Antagonist Protocol in Women Over 40 Years Undergoing ICSI Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Assistant professor of obstetrics and gynecology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/2021OBSGN 1
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Stimulation
MeSH Terms: interventions — Letrozole; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard GnRH antagonist protocol (Active Comparator): Gonadotropins (300-450 IU) IM start on cycle day 2 then the dose modulated according to response
  Interventions: Drug: Letrozole 2.5mg tablet
- Aromatase inhibitor/flexible antagonist protocol (Active Comparator): letrozole orally in a dose of 2.5 mg daily, on day 2 of cycle for 5 days and gonadotropins (300-450 IU) IM start on cycle day 3. then the dose modulated according to response
  Interventions: Drug: Letrozole 2.5mg tablet

INTERVENTIONS:
Drug: Letrozole 2.5mg tablet — letrozole (femara, Novartis) orally in a dose of 2.5 mg daily, on day 2 of cycle for 5 days and gonadotropins (300-450 IU) IM start on cycle day 3. then the dose modulated according to response
  Other Names: Gonadotropins units

SUMMARY:
The aim of this study To compare the clinical and laboratory outcomes of two ovarian stimulation protocols (standard GnRH antagonist protocol and aromatase inhibitor/ antagonist protocol) in women (40-44) years undergoing ICSI cycle.

DETAILED DESCRIPTION:
Fertility is known to decline significantly in women after the age of 35 years, and fecundity is almost completely lost after the age of 45 . As age increases the natural fecundity and pregnancy rates after assisted reproduction decrease .This reduction in fecundity is thought to be due to ovarian aging mainly, which is defined as a decline in both the quantity and quality of the ovarian follicle pool .The increase in patient's age is associated with poor ovarian response, as represented by smaller ovarian volume, lower antral follicle count and poor stromal vascularity. In addition to the reduction in fecundity, there is an increase in spontaneous abortion rates in this group of women .It has been reported that about 19% of all women undergo ART are 40 years, and they could be considered as expected poor responders .Various protocols of ovarian stimulation have been proposed to optimize IVF results in this age group, however, satisfactory results remain a challenge . The lack of initial central down-regulation in early follicular phase and adequate prevention of premature luteinizing hormone (LH) surge in late follicular phase provide GnRH antagonist protocol as a potentially proper option .The use of aromatase inhibitors in a GnRH antagonist protocol was suggested by some studies [Mit. Yarali and colleagues demonstrated that adjuvant therapy with letrozole could improve the response [Yarali et al., 2009]. Meanwhile, in another study, adding letrozole to ovarian stimulation has no positive effect on the likelihood of pregnancy . Letrozole is a selective, non-steroidal third generation aromatase inhibitor. Letrozole causes a reduction in conversion of androstenedione and testosterone to estrone and estradiol by inhibiting the aromatase enzyme activity . According to some published studies, the decline in early follicular phase estrogen levels, and consequently decrease in negative feedback of estrogen on FSH release in hypothalamic-pituitary axis cause an increase in endogenous gonadotropin secretion and stimulation of ovarian follicular growth. In addition, an increase in intraovarian androgens secondary to aromatase inhibition, augments the follicular sensitivity to FSH stimulation and follicular growth . Letrozole has no antiestrogenic effect over the endometrium . These reports prompted us to hypothesize that use of letrozole as a co-treatment agent in GnRH antagonist protocol might enhance cycle outcomes.

I

ELIGIBILITY:
Inclusion Criteria:

* Women between 40- 44-years undergoing ICSI cycle with FSH less than 15 and AMH more than 0.30.

Exclusion Criteria:

* Azoospermia in male partner,
* Previous ovarian surgery,
* Severe endometriosis,
* Uterine cavity lesion
* Metabolic or endocrine disorders including hyperprolactinemia and ypo/hyperthyroidism.
* Previous failed ICSI cycle.
* BMI more than 30.

Ages: 40 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
live birth rate | 1 year after embryo transfer
  deliveries ≥22 weeks gestation with heartbeat and breath

SECONDARY OUTCOMES:
positive hCG | 2 weeks after FET
  serum β-hCG ≥10 mIU/mL
clinical pregnancy | 5 weeks' gestation
  presence of intrauterine gestational sac by trans-vaginal ultrasound at gestational weeks.
Total gonadotropin /cycle (IU), | two weeks
  number of gonadotropin units needed per cycle
Duration of stimulation (Day), | two weeks
  number of days needed for stimulation
Endometrial thickness (mm) | two weeks
  measure endometrial thickness
serum E2 levels | two weeks
  measuring E2 level during stimulation
Follicles number | two weeks
  number of follicles during stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No